CLINICAL TRIAL: NCT03496766
Title: An Open Label Phase II Study of Tipifarnib in Advanced Squamous Non-small Cell Lung Cancer With HRAS Mutations
Brief Title: Tipifarnib in Advanced Squamous NSCLC With Oncogen HRAS MutAtionS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The recruitment was closed prematurely to due to slow recruitment.
Sponsor: Spanish Lung Cancer Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GECP17/04_THOMAS; 2017-004822-13 (EudraCT Number); KO-IST-003 (Other: KURA Oncology)
Record Dates: First submitted 2018-03-13; First posted 2018-04-12 (Actual); Results first posted 2024-03-29 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tipifarnib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): Tipifarnib 600 mg, po, bid daily on days 1-7 and 15-21 of 28-day treatment cycles for up to 24 months
  Interventions: Drug: Tipifarnib

INTERVENTIONS:
Drug: Tipifarnib — Tipifarnib 600 mg will be administered until progression
  Other Names: Zarnestra

SUMMARY:
This Phase II study consists of 2 parts: 1) pre-screening phase and 2) treatment phase.

The pre-screening phase will investigate the presence of HRAS mutations in subjects with a histologically or cytologically confirmed diagnosis of squamous non-small cell lung cancer (SQ-NSCLC). Subjects may participate in the pre-screening phase at initial diagnosis or following prior lines of therapy for SQ-NSCLC.

The treatment phase will investigate the antitumor activity in terms of ORR of tipifarnib in subjects with locally advanced squamous non-small cell lung cancer (SQ-NSCLC) with HRAS mutations and for whom there is no curative therapy available.

DETAILED DESCRIPTION:
Subject enrolment may proceed with information available on tumor HRAS status previously generated during the pre-screening phase, but all subjects must consent to provide tumor slides (or tumor tissue block) from a prior diagnostic biopsy for a retrospective testing of RAS gene status, including T81C polymorphism, and other potential biomarkers at a central facility.

Tipifarnib will be administered at a starting dose of 600 mg, po, bid daily on days 1-7 and 15-21 of 28-day treatment cycles. In the absence of unmanageable toxicities, subjects may continue to receive tipifarnib treatment for up to 24 months in the absence of disease progression and unmanageable toxicity. Treatment may continue beyond 24 months if there is documented evidence of continued clinical benefit.

Tumor assessments will be performed at screening and approximately every 8 weeks for the first 6 months (cycles 2, 4, 6) and then every 12 weeks (cycles 9, 12, 15, etc.) until disease progression, starting at the end of Cycle 2. Additional tumor assessments may be conducted if deemed necessary by the Investigator or for a confirmation of an objective response. Subjects who discontinue tipifarnib treatment for reasons other than disease progression must continue tumor assessments until disease progression, withdrawal of subject's consent to study procedures or initiation of another anticancer therapy.

Determination of objective tumor response will be performed by the Investigator according to the Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1. Electronic copies of tumor images may be de-identified of subject's personal information at the clinical sites and collected by the Sponsor to undergo an external independent radiological review if the sponsor deems it necessary for the final assessment of treatment efficacy. Subjects with a solitary site of disease who have experienced a response may be considered for surgical resection. Subjects with a best response of a partial response and residual disease after salvage surgery will be eligible to continue on study therapy. Information on the duration of response to the last prior therapy will be collected.

Upon disease progression, subjects will be followed approximately every 12 weeks for survival until either death or 24 months after accrual in the subject's study cohort has been completed, whichever occurs first. Information on subsequent anticancer therapy will be collected.

All subjects will be followed-up for safety during treatment and for approximately 30 additional days after treatment discontinuation (or until immediately before the administration of another anticancer treatment). Additional safety follow up may be conducted if unresolved toxicity is present at the End of Treatment visit.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a histologically or cytologically confirmed diagnosis of squamous non-small cell lung cancer (SQ-NSCLC) for which there is no curative therapy available.
2. Subject has relapsed (progressive disease) or is refractory to one or more prior therapies. In the case of therapy received in the adjuvant or neo-adjuvant setting, relapse must have occurred within 12 months to be considered prior therapy. Subject may have received prior immunotherapy.
3. Subject has a tumor that carries a missense HRAS mutation. HRAS status may have been assessed either in blood, primary tumor tissue, recurrent or metastatic disease.
4. Subject has consented to provide tumor slides (or tumor tissue blocks) for biomarker evaluation. Before enrolment the site must confirm the availability of the tumor sample. If there is no sample available, the trial chair must be contacted for approval. If enrolment in the treatment portion of the study has taken place based on HRAS mutant status as assessed using a blood sample, tumor tissue must be sent before starting cycle 2 of treatment, and It will be used in part for confirmation of HRAS mutant tumor status. Confirmation of HRAS mutant status in tumor tissue is required for continuation of treatment. If HRAS mutation is not confirmed in tumor but is clearly positive in blood, the trial chair will be contacted for approval and the treatment could be maintained. All treated subjects will be evaluated for safety.

6. At least 2 weeks since the last systemic therapy regimen prior to enrolment. Subjects must have recovered to NCI CTCAE v. 4.03 < Grade 2 from all acute toxicities (excluding Grade 2 toxicities that are not considered a safety risk by the Sponsor and Investigator) or toxicity must be deemed irreversible by the Investigator.

7. At least 2 weeks since last radiotherapy. If radiation was localized to the only site of measurable disease, there must be documentation of disease progression of the irradiated site. Subjects must have recovered from all acute toxicities from radiotherapy. Subjects may be on a daily dose of corticosteroids (≤ 20mg prednisone or equivalent), as part of their management from prior radiotherapy.

8. ECOG (Eastern cooperative oncology group) performance status of 0 or 1. 9. Acceptable liver function:

1. Bilirubin less than 1.5 times upper limit of normal (x ULN); does not apply to subjects with Gilbert's syndrome diagnosed as per institutional guidelines.
2. AST Aspartate Amino-transferasa (SGOT) and ALT Aspartate-Alanina-transferase (SGPT) less than 3 x ULN; if liver metastases are present, then ≥ 5 x ULN is allowed.

   10. Acceptable renal function with serum creatinine less than 1.5 x ULN or a calculated creatinine clearance ≥ 60 mL/min using the Cockcroft-Gault formula.

   11. Acceptable hematologic status:

a. ANC (absolut neuthophil count) ≥ 1000 cells/μL. b. Platelet count ≥ 75,000/μL. c. Hemoglobin ≥ 9.0 g/dL. 12. Female subjects must be either:

1. Of non-child-bearing potential (surgically sterilized or at least 2 years post-menopausal); or
2. If of child-bearing potential, subject must use an adequate method of contraception consisting of two-barrier method or one barrier method with a spermicide or intrauterine device. Both females and male subjects with female partners of child-bearing potential must agree to use an adequate method of contraception for 2 weeks prior to screening, during, and at least 4 weeks after last dose of trial medication. Female subjects must have a negative serum or urine pregnancy test within 72 hours prior to start of trial medication.
3. Not breast feeding at any time during the study. 13. Written and voluntary informed consent for the treatment phase understood, signed and dated.

Exclusion Criteria:

1. Ongoing treatment with an anticancer agent not contemplated in this protocol.
2. Prior treatment (at least 1 full treatment cycle) with an FTase inhibitor.
3. Any history of clinically relevant coronary artery disease or myocardial infarction within the last 3 years, New York Heart Association (NYHA) grade III or greater congestive heart failure, cerebro-vascular attack within the prior year, or current serious cardiac arrhythmia requiring medication except atrial fibrillation.
4. Known uncontrolled brain, leptomeningeal or epidural metastases (unless treated and well controlled for at least 4 weeks prior to Cycle 1 Day 1).
5. Non-tolerable > Grade 2 neuropathy or evidence of emerging or rapidly progressing neurological symptoms within 4 weeks of Cycle 1 Day 1. Non-tolerable grade 2 toxicities are defined as those with moderate symptoms that the patient is not able to endure for the conduct of instrumental activities of daily life or that persists ≥ 7 days.
6. Major surgery, other than diagnostic surgery, within 4 weeks prior to Cycle 1 Day 1, without complete recovery.
7. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy. Known infection with HIV, or an active infection with hepatitis B or hepatitis C.
8. Subjects who have exhibited allergic reactions to tipifarnib or structural compounds similar to tipifarnib or to the drug product excipients. This includes hypersensitivity to imidazoles, such as clotrimazole, ketoconazole, miconazole and others in this drug class. Patients with hypersensitivity to these agents will be excluded from enrolment.
9. Required use of concomitant medications classified as strong inhibitors or inducers of cytochrome P450 3A4 (CYP3A4) or UDP-glucuronosyltransferase (UGT)
10. Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the Investigator, pose an unacceptable risk to the subject in this study.
11. The subject has legal incapacity or limited legal capacity.
12. Significantly altered mental status that would limit the understanding or rendering of informed consent and compliance with the requirements of this protocol. Unwillingness or inability to comply with the study protocol for any reason.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis Paz Ares, MD, Study Chair — Hospital 12 de Octubre
Locations (30):
- Spain (30):
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, A Coruña
  - Hospital Virgen de los Lirios, Alcoy, Alicante
  - Hospital General Universitario de Elche, Elche, Alicante
  - ICO-Badalona, Badalona, Barcelona
  - ICO-Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Provincial de Castellón, Castellon, Castelló
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Universitario de la Arrixaca, El Palmar, Murcia
  - Hospital Costa del Sol, Marbella, Málaga
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Sant Joan de Reus, Reus, Tarragona
  - H. Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - H.U.Vall D´Hebrón, Barcelona
  - H. Clinic i Provincial, Barcelona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario de Ciudad Real, Ciudad Real
  - ICO Girona -H. Dr. Josep Trueta, Girona
  - Hospital de Jaén, Jaén
  - Hospital Lucus Agustí, Lugo
  - Hospital La Princesa, Madrid
  - Hospital Puerta de Hierro, Madrid
  - H. 12 de Octubre, Madrid
  - H. Carlos Haya, Málaga
  - H. Son Llàtzer, Palma de Mallorca
  - Hospital Clinico de Salamanca, Salamanca
  - Hospital Virgen de La Macrena, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - H. General U. de Valencia, Valencia
  - Hospital La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Web page of the sponsor where users can find more information about Fundación GECP studies — http://www.gecp.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Arm
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental Arm
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Spain | 9
Cigarette Smoking History [Count of Participants; unit: Participants]
  Never smoker (<= 100 cigarettes/lifetime) | 0
  Former smoker (>= 1 year) | 5
  Active smoker | 4
ECOG Performance status [Count of Participants; unit: Participants] — ECOG Performance Status Scale: It describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability
  GRADES:
  ECOG 0: Fully active. ECOG 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature ECOG 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours ECOG 3: Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours ECOG 4: Completely disabled
  Participants
    ECOG 0 | 0
    ECOG 1 | 9
    ECOG 2 | 0
    ECOG 3 | 0
    ECOG 4 | 0
Pulse rate [Mean (Standard Deviation); unit: bpm] | 88.8 (12.1)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 121.8 (22.2)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 73.2 (10.4)
Clinical Stage at inclusion [Count of Participants; unit: Participants] — Staging is a classification where cancer is located, if or where it has spread and whether it's affecting other parts of the body.
  * Stage IIIB. The primary tumor is 5cm or smaller and cancer has spread to lymph nodes
  * Stage IIIC. The tumor may be any size and cancer has spread to lymph nodes, cannot be removed with surgery
  * Stage IVA cancer has spread within the chest and/or has spread to 1 area outside of the chest.
  * Stage IVB has spread outside of the chest to more than 1 place in 1 organ or to more than 1 organ. This is considered a worse outcome
  Participants
    IIIB-IIIC | 1
    IVA | 4
    IVB | 4
Prior Therapy Best Response [Count of Participants; unit: Participants] — Best Response will be evaluated in this trial using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee (v.1.1).
  Evaluation of Target Lesions Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient PD
  Participants
    Partial Response | 3
    Stable Disease | 4
    Progression Disease | 2
Antineoplastic TMT Chemotherapy First Line [Count of Participants; unit: Participants]
  Carboplatin | 1
  Cisplatin | 2
  Cisplatin + Gemcitabine | 1
  Paclitaxel | 1
  Pembrolizumab | 3
  Carboplatin + Pemetrexed + Pembrolizumab | 1
Antineoplastic TMT Chemotherapy Second Line [Count of Participants; unit: Participants] — Population: One subject didn't receive 2nd line of antineoplastic treatment
  Participants
    number analyzed (Participants) | 8
    Carboplatin | 1
    Carboplatin + Gemcitabine | 1
    Carboplatin + Vinorebine | 1
    Cisplatin + Gemcitabine | 1
    Gemcitabine | 1
    Paclitaxel | 2
    Pembrolizumab + Radium 223 | 1
Antineoplastic TMT Chemotherapy Third Line [Count of Participants; unit: Participants] — Population: 6 subject didn't receive 3rd line of antineoplastic treatment
  Participants
    number analyzed (Participants) | 3
    Carboplatin | 1
    Cetuximab | 1
    Docetaxel | 1
Antineoplastic TMT Chemotherapy Fourth Line [Count of Participants; unit: Participants] — Population: 7 subject didn't receive 4 line of antineoplastic treatment
  Participants
    number analyzed (Participants) | 2
    Avelumab | 1
    Nivolumab | 1
Antineoplastic TMT Chemotherapy Fifth Line [Count of Participants; unit: Participants] — Population: 7 subject didn't receive 5th line of antineoplastic treatment
  Participants
    number analyzed (Participants) | 2
    Docetaxel | 1
    Etoposide | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response
Description: To determine the antitumor activity in terms of objective response rate (ORR) of tipifarnib in subjects with locally advanced unresectable or metastatic, relapsed and/or refractory, squamous non-small cell lung cancer (SQ-NSCLC) with HRAS mutations.
  Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. Progressive disease (PD): at least a 20% increase in the sum of diameters of target lesions.
Time Frame: From the first dose until progression disease, assessed from the first dose until the first assessment at week 6 from the first dose
Population: Per protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm
Number analyzed (Participants) | 6
Participants
  Stable Disease | 2
  Progression Disease | 4

2. Secondary Outcome: Progression Free Survival
Description: Defined as the time from the start date of treatment TMT as the origin of follow-up and the first progression or death as final date.
Time Frame: From the start of treatment until first progression or death.
Measure: Median (Standard Deviation); unit: months
Arm/Group | Experimental Arm
Number analyzed (Participants) | 9
months | 8.6 (18.7)

3. Secondary Outcome: Overall Survival
Description: Defined as the length of time from either the date of diagnosis or the start of the treatment that patients diagnosed with the disease are still alive.
Time Frame: From the date of randomization until end of follow up,up to 24 months
Measure: Median (Full Range); unit: Months
Arm/Group | Experimental Arm
Number analyzed (Participants) | 9
Months | 12.4 [9.7 to 21.7]

ADVERSE EVENTS:
Time Frame: 25 months
Description: The severity of AE will be determined using CTCA version 4
Arm/Group | Experimental Arm
All-Cause Mortality (participants affected / at risk) | 9/9
Serious Adverse Events (participants affected / at risk) | 9/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm (N=9)
Renal and urinary disorders (Renal and urinary disorders) | 6 (6)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Platelet count decreased (Blood and lymphatic system disorders) | 2 (2)
Nervous system disorders (Nervous system disorders) | 1 (1)
Thromboembolic event (Blood and lymphatic system disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm (N=9)
Anemia (Blood and lymphatic system disorders) | 9 (9)
Hyperglycemia (Investigations) | 7 (7)
Confusion (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The recruitment was closed prematurely to due to slow recruitment, so there are no consistent data to achieve any relevant conclusion at this point.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-15): https://cdn.clinicaltrials.gov/large-docs/66/NCT03496766/Prot_SAP_000.pdf